CLINICAL TRIAL: NCT03651635
Title: To Assess and Validate the Use of MR-proADM and the CT-proET-1/MR-proADM Ratio as Prognostic Markers During the First 7 Days of ICU Treat-ment
Brief Title: MR-proADM and CT-proET-1 During ICU Treatment
Acronym: MR-proADM
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: ThermoFisher Scientific Brahms Biomarkers France (Industry)
Responsible Party: Sponsor
Other Study IDs: proADM
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Acute Phase Biomarkers; Medical ICU Admitted Patients
Keywords: ICU; Biomarkers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the process of the study we will collect at most 8 additional blood samples (3ml each). The collection of the blood samples will be paired with routine laboratory checks. All other parameters (health related personal data, comorbidities, values of hemodynamic will be reviewed from the chart or evaluated in line with routine daily investigations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical ICU Patients: All patients admitted to the medical intensive care unit of the University hospital of Zurich during the recruitment period
  Interventions: Diagnostic Test: Blood sampling for MR-proADM & CT-proET-1

INTERVENTIONS:
Diagnostic Test: Blood sampling for MR-proADM & CT-proET-1 — Collection of at most 8 blood samples (3ml each) per Patient admitted to the study and sampling for MR-proADM & CT-proET-1

SUMMARY:
This pilot-study will be a prospective, single-centre, observational study including 100 critically ill patients consecutively admitted to the medical intensive care unit (ICU) of the University hospital of Zurich, Switzerland, to assess and validate the use of MR-proADM and the CT-proET1/MR-proADM-ratio as prognostic markers in critically ill patients.

DETAILED DESCRIPTION:
This pilot-study will be a prospective, single-centre, observational study including 100 critically ill patients consecutively admitted to the medical intensive care unit (ICU) of the University hospital of Zurich, Switzerland, to assess and validate the use of MR-proADM and the CT-proET1/MR-proADM-ratio as prognostic markers in critically ill patients. After obtaining informed consent of the patient or approval of a legal representative and meeting of the inclusion, as well as missing exclusion criteria the patients will be enrolled.

At study enrolment patient health status will be assessed by health related diagnosis and the Charlson comorbidity index. This information is obtained routinely in every patient in our ICU. The Charlson comorbidity index is calculated based on the medical history of the patient. The values of MR-proADM and CT-proET-1 will be measured daily over the first 7 days of the ICU stay. If a patient is discharged before day 7, no further measurements will be performed. The blood samples will be collected together with the routine blood check on admission, as well as each morning. Clinical evaluation of the patients will take place each morning including the evaluation of the hemodynamics, organ dysfunction, microcirculation and the need for vasopressors.

The severity of illness of the patient will be assessed using the SAPS II score and the SOFA score. SAPS-II reflects the physiological status of the patient within the first 24 hours (admission severity) and the SOFA score the number of failing organs (respiration, coagulation, liver, cardiovascular, CNS, renal). The SAPS-II will be assessed on Visit 3 and the SOFA daily using the information obtained during the routine clinical examination and the laboratory results of the day. SAPS II and SOFA scores are part of the routine assessment of all our patients in the ICU and are used as quality indicators.

The status of the microcirculation is assessed using clinical signs (mottling score, capillary refill time and sublingual microcirculation functional status) and laboratory parameters reflecting the degree of tissue oxygen extraction such as SaO2-SvO2 gap, Pv-aCO2 gap and the arterial lactate concentration. All these parameters are delivered by the blood gas analyser located in the ICU from an arterial and a venous blood sample of 1.5 ml each drawn via the arterial and central venous line respectively. These catheters and blood samples are part of the routine hemo-dynamic monitoring and assessment of the critically ill patient in our ICU.

The patients' survival status will be assessed on day 7 and day 28 after study enrolment. In addition, ICU and hospital mortality are recorded. If the patient is still in the hospital on day 28, survival data will be taken from the medical record. In the case the patient is dismissed from the hospital the study team will contact him by phone call. If he is not reachable (documented attempts) the study team will contact his general practitioner. To be in line with data protection requirements the patient gives the consent to contact the general practitioner in the informed consent form. No other information than the survival status will be collected at this stage. Data collection for the study ends 28 (± 3 days) days after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the medical intensive care unit of the University hospital of Zurich during the recruitment period
* Male and female participants ≥ 18 years
* Written informed consent by the participant after information about the research project or if the patient is incapable of giving informed consent, a legal representative has confirmed the presumed will of the participant (according Art. 15 KlinV emergency patients)

Exclusion Criteria:

* Inability of the conscious patients to follow the experimental procedure, e.g. because of insufficient language skills (German), mental illness, dementia etc.
* Pregnancy
* Participation in ongoing clinical trials of other departments of the University Hospital Zurich

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the medical intensive care unit of the University hospital of Zurich during the recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUROCCs) for MR-proADM | 7 days
  Area under the concentration-time curve (AUROCCs) over 7 days for MR-proADM grouped by SOFA-Score ≥ 7 on day 7
Area under the concentration-time curve (AUROCCs) for the CT-proET-1/MR-proADM-ratio | 7 days
  Area-under the concentration-time-curve (AUROCCs) over 7 days for the CT-proET-1/MR-proADM-ratio grouped by SOFA-Score ≥ 7 on day 7

SECONDARY OUTCOMES:
Correlation between area under the concentration-time curve for MR-proADM and microcirculation status | 7 days
  Correlation between area under the concentration-time curve for MR-proADM and microcirculation status (mottling score, capillary refill time, sublingual microcirculation functional status) on day 7
Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and microcirculation status | 7 days
  Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and microcirculation status (mottling score, capillary refill time, sublingual microcirculation functional status) on day 7
Correlation between area under the concentration-time curve for MR-proADM and cardiac biomarkers | 7 days
  Correlation between area under the concentration-time curve for MR-proADM and cardiac biomarkers (NT-proBNP, Troponin T) during the first 7 days of ICU stay
Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and cardiac biomarkers | 7 days
  Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and cardiac biomarkers (NT-proBNP, Troponin T) during the first 7 days of ICU stay
Correlation between area under the concentration-time curve for MR-proADM and biomarkers of inflammation | 7 days
  Correlation between area under the concentration-time curve for MR-proADM and biomarkers of inflammation (C-reactive protein, procalcitonin, interleukin-6) during the first 7 days of ICU stay
Correlation between area under the concentration-time curve for the CT-proET-1/MR-proADM-ratio and biomarkers of inflammation | 7 days
  Correlation between area under the concentration-time curve for the CT-proET-1/MR-proADM-ratio and biomarkers of inflammation (C-reactive protein, procalcitonin, interleukin-6) during the first 7 days of ICU stay
Correlation between area under the concentration-time curve for MR-proADM and renal dysfunction | 7 days
  Correlation between area under the concentration-time curve for MR-proADM and renal dysfunction (AKI defined by KDIGO-Classification) on day 7 or ICU discharge
Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and renal dysfunction | 7 days
  Correlation between area under the concentration-time curve for the CT-proET1/MR-proADM-ratio and renal dysfunction (AKI defined by KDIGO-Classification) on day 7 or ICU discharge
Admission plasma levels of MR-proADM as a predictor of multiorgan dysfunction | 7 days
  Admission plasma levels of MR-proADM as a predictor of multiorgan dysfunction (SOFA-Score ≥ 7) on day 7 of ICU treatment (ROC-AUC)
Admission plasma levels of the CT-proET1/MR-proADM-ratio as a predictor of multiorgan dysfunction | 7 days
  Admission plasma levels of the CT-proET1/MR-proADM-ratio as a predictor of multiorgan dysfunction (SOFA-Score ≥ 7) on day 7 of ICU treatment (ROC-AUC)
AUROCCs for MR-proADM during the first 7 days of ICU treatment as predictors of mortality | 28 days
  AUROCCs for MR-proADM during the first 7 days of ICU treatment as predictors of mortality on day 7, 28 and hospital-mortality
AUROCCs for the MR-proADM/CT-proET-1-ratio during the first 7 days of ICU treatment as predictors of mortality | 28 days
  AUROCCs for the MR-proADM/CT-proET-1-ratio during the first 7 days of ICU treatment as predictors of mortality on day 7, 28 and hospital-mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, MD, Principal Investigator — University Zürich/ University Hospital Zürich
Locations (1):
- University Hospital Zurich, Medical intensive care unit, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espana PP, Capelastegui A, Quintana JM, Bilbao A, Diez R, Pascual S, Esteban C, Zalacain R, Menendez R, Torres A. Validation and comparison of SCAP as a predictive score for identifying low-risk patients in community-acquired pneumonia. J Infect. 2010 Feb;60(2):106-13. doi: 10.1016/j.jinf.2009.11.013. Epub 2009 Dec 2. PMID 19961875
- [Background] Fine MJ, Auble TE, Yealy DM, Hanusa BH, Weissfeld LA, Singer DE, Coley CM, Marrie TJ, Kapoor WN. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997 Jan 23;336(4):243-50. doi: 10.1056/NEJM199701233360402. PMID 8995086
- [Background] Lim WS, van der Eerden MM, Laing R, Boersma WG, Karalus N, Town GI, Lewis SA, Macfarlane JT. Defining community acquired pneumonia severity on presentation to hospital: an international derivation and validation study. Thorax. 2003 May;58(5):377-82. doi: 10.1136/thorax.58.5.377. PMID 12728155
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Pierrakos C, Vincent JL. Sepsis biomarkers: a review. Crit Care. 2010;14(1):R15. doi: 10.1186/cc8872. Epub 2010 Feb 9. PMID 20144219
- [Background] Hinson JP, Kapas S, Smith DM. Adrenomedullin, a multifunctional regulatory peptide. Endocr Rev. 2000 Apr;21(2):138-67. doi: 10.1210/edrv.21.2.0396. PMID 10782362
- [Background] Eto T. A review of the biological properties and clinical implications of adrenomedullin and proadrenomedullin N-terminal 20 peptide (PAMP), hypotensive and vasodilating peptides. Peptides. 2001 Nov;22(11):1693-711. doi: 10.1016/s0196-9781(01)00513-7. PMID 11754955
- [Background] Morgenthaler NG, Struck J, Alonso C, Bergmann A. Measurement of midregional proadrenomedullin in plasma with an immunoluminometric assay. Clin Chem. 2005 Oct;51(10):1823-9. doi: 10.1373/clinchem.2005.051110. Epub 2005 Aug 11. PMID 16099941
- [Background] Papassotiriou J, Morgenthaler NG, Struck J, Alonso C, Bergmann A. Immunoluminometric assay for measurement of the C-terminal endothelin-1 precursor fragment in human plasma. Clin Chem. 2006 Jun;52(6):1144-51. doi: 10.1373/clinchem.2005.065581. Epub 2006 Apr 20. PMID 16627560
- [Background] Albrich WC, Dusemund F, Ruegger K, Christ-Crain M, Zimmerli W, Bregenzer T, Irani S, Buergi U, Reutlinger B, Mueller B, Schuetz P. Enhancement of CURB65 score with proadrenomedullin (CURB65-A) for outcome prediction in lower respiratory tract infections: derivation of a clinical algorithm. BMC Infect Dis. 2011 May 3;11:112. doi: 10.1186/1471-2334-11-112. PMID 21539743
- [Background] Albrich WC, Ruegger K, Dusemund F, Schuetz P, Arici B, Litke A, Blum CA, Bossart R, Regez K, Schild U, Guglielmetti M, Conca A, Schafer P, Schubert M, de Geest S, Reutlinger B, Irani S, Burgi U, Huber A, Muller B. Biomarker-enhanced triage in respiratory infections: a proof-of-concept feasibility trial. Eur Respir J. 2013 Oct;42(4):1064-75. doi: 10.1183/09031936.00113612. Epub 2013 Jan 24. PMID 23349444
- [Background] Bello S, Lasierra AB, Minchole E, Fandos S, Ruiz MA, Vera E, de Pablo F, Ferrer M, Menendez R, Torres A. Prognostic power of proadrenomedullin in community-acquired pneumonia is independent of aetiology. Eur Respir J. 2012 May;39(5):1144-55. doi: 10.1183/09031936.00080411. Epub 2011 Nov 10. PMID 22075489
- [Background] Christ-Crain M, Morgenthaler NG, Stolz D, Muller C, Bingisser R, Harbarth S, Tamm M, Struck J, Bergmann A, Muller B. Pro-adrenomedullin to predict severity and outcome in community-acquired pneumonia [ISRCTN04176397]. Crit Care. 2006;10(3):R96. doi: 10.1186/cc4955. Epub 2006 Jun 28. PMID 16805922
- [Background] Christ-Crain M, Morgenthaler NG, Struck J, Harbarth S, Bergmann A, Muller B. Mid-regional pro-adrenomedullin as a prognostic marker in sepsis: an observational study. Crit Care. 2005;9(6):R816-24. doi: 10.1186/cc3885. Epub 2005 Nov 15. PMID 16356231
- [Background] Courtais C, Kuster N, Dupuy AM, Folschveiller M, Jreige R, Bargnoux AS, Guiot J, Lefebvre S, Cristol JP, Sebbane M. Proadrenomedullin, a useful tool for risk stratification in high Pneumonia Severity Index score community acquired pneumonia. Am J Emerg Med. 2013 Jan;31(1):215-21. doi: 10.1016/j.ajem.2012.07.017. Epub 2012 Sep 20. PMID 23000327
- [Background] Daka B, Olausson J, Larsson CA, Hellgren MI, Rastam L, Jansson PA, Lindblad U. Circulating concentrations of endothelin-1 predict coronary heart disease in women but not in men: a longitudinal observational study in the Vara-Skovde Cohort. BMC Cardiovasc Disord. 2015 Nov 14;15:146. doi: 10.1186/s12872-015-0141-y. PMID 26573599
- [Background] Guignant C, Voirin N, Venet F, Lepape A, Monneret G. Persistent high level of circulating midregional-proadrenomedullin and increased risk of nosocomial infections after septic shock. J Trauma Acute Care Surg. 2012 Jan;72(1):293-6. doi: 10.1097/TA.0b013e31823a0d23. PMID 22310138
- [Background] Huang DT, Angus DC, Kellum JA, Pugh NA, Weissfeld LA, Struck J, Delude RL, Rosengart MR, Yealy DM. Midregional proadrenomedullin as a prognostic tool in community-acquired pneumonia. Chest. 2009 Sep;136(3):823-831. doi: 10.1378/chest.08-1981. Epub 2009 Apr 10. PMID 19363212
- [Background] Liu D, Xie L, Zhao H, Liu X, Cao J. Prognostic value of mid-regional pro-adrenomedullin (MR-proADM) in patients with community-acquired pneumonia: a systematic review and meta-analysis. BMC Infect Dis. 2016 May 26;16:232. doi: 10.1186/s12879-016-1566-3. PMID 27230573
- [Background] Lundberg OH, Bergenzaun L, Ryden J, Rosenqvist M, Melander O, Chew MS. Adrenomedullin and endothelin-1 are associated with myocardial injury and death in septic shock patients. Crit Care. 2016 Jun 9;20(1):178. doi: 10.1186/s13054-016-1361-y. PMID 27282767
- [Background] Schuetz P, Christ-Crain M, Morgenthaler NG, Struck J, Bergmann A, Muller B. Circulating precursor levels of endothelin-1 and adrenomedullin, two endothelium-derived, counteracting substances, in sepsis. Endothelium. 2007 Nov-Dec;14(6):345-51. doi: 10.1080/10623320701678326. PMID 18080871
- [Background] Schuetz P, Christ-Crain M, Zimmerli W, Mueller B. Repeated measurements of endothelin-1 precursor peptides predict the outcome in community-acquired pneumonia. Intensive Care Med. 2011 Jun;37(6):970-80. doi: 10.1007/s00134-011-2208-2. Epub 2011 Mar 11. PMID 21394616
- [Background] Schuetz P, Stolz D, Mueller B, Morgenthaler NG, Struck J, Mueller C, Bingisser R, Tamm M, Christ-Crain M. Endothelin-1 precursor peptides correlate with severity of disease and outcome in patients with community acquired pneumonia. BMC Infect Dis. 2008 Feb 28;8:22. doi: 10.1186/1471-2334-8-22. PMID 18304365
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Champion HR, Sacco WJ, Carnazzo AJ, Copes W, Fouty WJ. Trauma score. Crit Care Med. 1981 Sep;9(9):672-6. doi: 10.1097/00003246-198109000-00015. PMID 7273818
- [Background] Fleming S, Gill P, Jones C, Taylor JA, Van den Bruel A, Heneghan C, Thompson M. Validity and reliability of measurement of capillary refill time in children: a systematic review. Arch Dis Child. 2015 Mar;100(3):239-49. doi: 10.1136/archdischild-2014-307079. Epub 2014 Sep 26. PMID 25260515
- [Background] Ait-Oufella H, Bige N, Boelle PY, Pichereau C, Alves M, Bertinchamp R, Baudel JL, Galbois A, Maury E, Guidet B. Capillary refill time exploration during septic shock. Intensive Care Med. 2014 Jul;40(7):958-64. doi: 10.1007/s00134-014-3326-4. Epub 2014 May 9. PMID 24811942
- [Background] Ait-Oufella H, Lemoinne S, Boelle PY, Galbois A, Baudel JL, Lemant J, Joffre J, Margetis D, Guidet B, Maury E, Offenstadt G. Mottling score predicts survival in septic shock. Intensive Care Med. 2011 May;37(5):801-7. doi: 10.1007/s00134-011-2163-y. Epub 2011 Mar 4. PMID 21373821
- [Background] Coudroy R, Jamet A, Frat JP, Veinstein A, Chatellier D, Goudet V, Cabasson S, Thille AW, Robert R. Incidence and impact of skin mottling over the knee and its duration on outcome in critically ill patients. Intensive Care Med. 2015 Mar;41(3):452-9. doi: 10.1007/s00134-014-3600-5. Epub 2014 Dec 17. PMID 25516087
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Assink-de Jong E, de Lange DW, van Oers JA, Nijsten MW, Twisk JW, Beishuizen A. Stop Antibiotics on guidance of Procalcitonin Study (SAPS): a randomised prospective multicenter investigator-initiated trial to analyse whether daily measurements of procalcitonin versus a standard-of-care approach can safely shorten antibiotic duration in intensive care unit patients--calculated sample size: 1816 patients. BMC Infect Dis. 2013 Apr 16;13:178. doi: 10.1186/1471-2334-13-178. PMID 23590389
- [Background] Safdar N, Fine JP, Maki DG. Meta-analysis: methods for diagnosing intravascular device-related bloodstream infection. Ann Intern Med. 2005 Mar 15;142(6):451-66. doi: 10.7326/0003-4819-142-6-200503150-00011. PMID 15767623
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Pranskunas A, Koopmans M, Koetsier PM, Pilvinis V, Boerma EC. Microcirculatory blood flow as a tool to select ICU patients eligible for fluid therapy. Intensive Care Med. 2013 Apr;39(4):612-9. doi: 10.1007/s00134-012-2793-8. Epub 2012 Dec 20. PMID 23263029
- [Background] Trzeciak S, McCoy JV, Phillip Dellinger R, Arnold RC, Rizzuto M, Abate NL, Shapiro NI, Parrillo JE, Hollenberg SM; Microcirculatory Alterations in Resuscitation and Shock (MARS) investigators. Early increases in microcirculatory perfusion during protocol-directed resuscitation are associated with reduced multi-organ failure at 24 h in patients with sepsis. Intensive Care Med. 2008 Dec;34(12):2210-7. doi: 10.1007/s00134-008-1193-6. Epub 2008 Jul 2. PMID 18594793
- [Background] Hilty MP, Pichler J, Ergin B, Hefti U, Merz TM, Ince C, Maggiorini M. Assessment of endothelial cell function and physiological microcirculatory reserve by video microscopy using a topical acetylcholine and nitroglycerin challenge. Intensive Care Med Exp. 2017 Dec;5(1):26. doi: 10.1186/s40635-017-0139-0. Epub 2017 May 18. PMID 28523563